CLINICAL TRIAL: NCT02955108
Title: The Effect of Distractive Auditory Stimuli (Music) on Dyspnea and Anxiety During Exercise in Adults With Chronic Respiratory Disease
Brief Title: The Effect of Distractive Auditory Stimuli (Music) on Dyspnea and Anxiety During Exercise in Adults With Chronic Respiratory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-01676
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music first then no music (Experimental)
  Interventions: Procedure: Distractive Auditory Stimuli; Procedure: No Distractive Auditory Stimuli
- no music first then music (Experimental)
  Interventions: Procedure: Distractive Auditory Stimuli; Procedure: No Distractive Auditory Stimuli

INTERVENTIONS:
Procedure: Distractive Auditory Stimuli — Participants will self-select 1 music piece from a list of choices to keep the rhythm and tempo consistent throughout the 6MWT. The instructions to participants for selecting the music will be standardized. TThe music volume will be standardized to be "moderately loud" as rated by participants for the music condition. Participants will not be specifically instructed to synchronize their walking movements with the music tempo. The music is based on a cognitive therapy (distraction) strategy conceptual framework. Music will be played during the 6MWT (in-task) only.
Procedure: No Distractive Auditory Stimuli — Participants will wear headphones with no music playing

SUMMARY:
The objective of this study is to look at the effects of distractive auditory stimuli (DAS) on reducing dyspnea intensity and related anxiety and increasing exercise tolerance. Investigators hope that compared to a no-music control condition, that under a music condition participants with COPD will (a) demonstrate increased self-paced walk distance and enjoyment; (b) have less dyspnea intensity, (c) experience less dyspnea anxiety; (d) have less fatigue and state anxiety; and (e) higher maximum heart rate. The upbeat music with a tempo of 90 - 100 bpm (an average-to-moderate walking tempo) is expected to have distractive and performance enhancing effects in order to increase tolerance to dyspnea and exercise. The long-term goal of this study is to increase physical activity in adults with COPD and RLD by promoting dyspnea and fatigue management through use of distractive auditory stimuli in the form of music.

DETAILED DESCRIPTION:
This randomized clinical trial will use a cross-over design. The research will include two within-subject factors, music versus no music and time. Each subject will be randomized a single time to receive either music first then no music, or alternatively, no music first then music during two walk tests.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* aged 40 years or older, with physician-diagnosed COPD
* a flow volume loop with a FEV1/FVC of < 0.70 in the past 12 months

  * medically cleared to participate in NYULMC's pulmonary rehabilitation program.

Exclusion Criteria:

* Inability to exercise due to musculoskeletalor neurological dysfunction
* Inability to walk independently (unaided)
* deafness or severe hearing impairment requiring hearing aids
* mMRC score = 0 ("I only get breathlessness with strenuous exercise").

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Dyspnea Intensity (DI) | 60 Minutes
  Borg Breathlessness Scale. The Borg dyspnea scale is a single-item rating scale, ranging between 0, "nothing at all", and 10, "very, very severe (maximal)". Patients will be asked to rate their level of dyspnea during the walk test using the 10-point Borg scale after the 6MWT.64 Validity of the Borg scale for measuring dyspnea intensity has been shown.65

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Norweg, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States